CLINICAL TRIAL: NCT04065711
Title: Multi-Center Study of the Soliton Rapid Acoustic Pulse (RAP) Device for the Treatment of Cellulite
Brief Title: Study of the Soliton Rapid Acoustic Pulse (RAP) Device for the Treatment of Cellulite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soliton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-002
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Cellulite
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- RAP Treatment (Experimental): Each treatment area will receive 30-40 minutes (30-40 individual doses) of RAP treatment.
  Interventions: Device: Soliton's Rapid Acoustic Pulse (RAP)

INTERVENTIONS:
Device: Soliton's Rapid Acoustic Pulse (RAP) — Treatment for the temporary improvement in the appearance of cellulite.

SUMMARY:
To evaluate the safety, and efficacy of Soliton's Rapid Acoustic Pulse (RAP) device for the temporary improvement in the appearance of cellulite.

DETAILED DESCRIPTION:
Multi-site clinical study to evaluate the safety, efficacy and tolerability of Soliton's Rapid Acoustic Pulse (RAP) device fo the temporary improvement in the appearance of cellulite.

ELIGIBILITY:
Inclusion Criteria:

* Female ages 18-50 years
* Seeking treatment of cellulite in the thigh and/or buttock areas
* Area of severe cellulite on the thigh and/or buttock with an average simplified Cellulite Severity Scale at Baseline ≥ 4.0 (Table 2)
* Having at least one dimple, or ridge-depression, in the treatment area, with a depth of approximately 5 mm or greater.
* Stable weight nominally +/- 5% for at least the past 6 months.
* Body Mass Index (B.M.I.) is ≤ 30
* Participant will not have had invasive or energy based cellulite treatments (liposuction, subcision, RF, laser, ESWT, etc.) for the prior 12 months.
* Participant will not have used topical based cellulite treatments for prior 6 months and will not use during the trial.
* Will not undergo any other cellulite treatments for a period of 12 months following RAP treatment.
* Participant is willing to participate in study and adhere to follow-up schedule
* Participant is able to read and comprehend English
* Participant has completed the Informed Consent Form

Exclusion Criteria:

* Participant is unwilling to have research photos taken of treatment areas in the presence of Sponsor's researchers.
* Participant is unwilling to have RAP treatment provided in the presence of Sponsor's researchers.
* Participant is pregnant or planning to become pregnant during the duration of the study.
* Has atrophic scars, or has a history of atrophic scars or keloids.
* Tattoo or former tattoo at or near treatment area.
* Metal or plastic implants in the area of the treatment (vascular stent, or implants in the hips, knees, etc.).
* Active electronic implants such as pacemakers, defibrillators, cochlear implants, nerve/brain stimulators, drug pump, etc.
* Medical disorder that would hinder the wound healing or immune response (no blood disorder, inflammatory disease, etc.).
* History of coagulopathy(ies) and/or on anticoagulant medication.
* Skin disorders (skin infections or rashes, extensive scarring, psoriasis, etc.) in the treatment area.
* Current smoker.
* Any surgical procedure in the prior 3 months, or planned during the duration of the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is specific to females ages 18-50 years.
Enrollment: 67 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-08-26 (Actual)

PRIMARY OUTCOMES:
Procedure Safety- All treated participants are free from unexpected adverse events | 12 weeks
  The primary objective is to demonstrate freedom from unexpected adverse
  events (UAEs) and serious adverse events (SAEs) directly attributable to the RAP device or treatment.

SECONDARY OUTCOMES:
RAP treatment effectiveness | 12 weeks, 26 weeks and 52 weeks
  To demonstrate temporary improvement in the appearance of cellulite as determined by blinded independent physician assessment (IPA) correctly identifying the 12-week post-treatment photographs from randomly placed side-by-side comparison of before and after photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Capelli, MD, Study Director — Soliton, Inc.
Locations (4):
- United States (4):
  - Clear Dermatology and Aesthetics Center Investigate MD, Scottsdale, Arizona
  - Chicago Cosmetic Surgery & Dermatology, Chicago, Illinois
  - Capital Laser and Skin Care, Chevy Chase, Maryland
  - SkinCare Physicians, Chestnut Hill, Massachusetts

IPD SHARING:
Plan to Share IPD: No